CLINICAL TRIAL: NCT04751123
Title: Assessment of Wheelchair First and Last Seating Pressure and Posture and Wheelchair Satisfaction
Brief Title: Does Prolonged Sitting Pressure Affect Sitting Pressure, Flexibility and Discomfort?
Acronym: (wheelchair)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Erdeo, PHD, Necmettin Erbakan University
Other Study IDs: NecmettinNEU
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: E07.796.980; G11.427.695
Keywords: wheelchair; seating pressure; posture; life quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ntroduction: Pressure sores and postural changes are observed in wheelchair users due to long sitting. Depending on this situation, the quality of life and activity participation level of these individuals decrease.

Method: This study will be conducted between March 1 and June 30, 2021 in Necmettin Erbakan University, Meram Faculty of Medicine, Physical Therapy and Rehabilitation Polyclinic. With the hamstring and trunk flexibility sit-lie test, six sensors placed on the sitting pressure sitting cushion, daily life activity FIM, skill assessment tests will be applied for manual and wheelchair users. Wheelchair Satisfaction CHART and quality of life World Health Organization Quality of Life (Whool ) will be evaluated with.

Application: Patients coming to the center spend 20 minutes on MAT. After resting, FIM will be evaluated with the sit-and-lie test. Afterwards, the patient will be put in a wheelchair. The initial sitting pressure will be taken as soon as you sit in the wheelchair. And at that time, CHART and WHOOL will be completed by asking the patient.

Conclusion: In the light of these evaluations, the change in initial sitting pressure and posture over time will be examined.

DETAILED DESCRIPTION:
HH.3. Scope:

Which is about 12.29% of the population consists of disabled people in Turkey and the highest rate of disability It is known that physical disability (1). Having at least one wheelchair of approximately 75 million worldwide according to 2019 data plays a critical role in improving mobility (2). In fact, the wheelchair is one of the most widely used assistive technology tools to increase personal mobility and is a precondition for those with limited mobility to enjoy their human rights, live in dignity and become more productive members in their community. For many people, a well-designed and well-equipped wheelchair can be the right step for social inclusion (3). More than half of wheelchair users need assistance with using their wheelchairs and daily living activities (4). The literature investigating the factors affecting wheelchair use mainly consists of variables related to the environment and physical characteristics of wheelchair users (4). Correct selection and configuration of wheelchairs can increase mobility, effectiveness and participation (5).

While sitting comfort is associated with softness and support, lack of support, unbalanced pressure distribution, biomechanics and fatigue factors are associated with sitting discomfort. Anatomical factors can cause characteristic tissue loads that appear to be associated with tissue damage, discomfort, or axillary posture or movement modifications. Following excessive or prolonged tissue loading, cell death may lead to the development of superficial or deep compression wounds (6). A superficial pressure sore first affects the skin layers near the epidermal tissue and is typically associated with damaging friction and shear forces with the presence of moisture and heat (7). Deep compression sores typically begin with the deformation of deep muscle and fat tissues beneath the ischial tuberocytes in the sitting position (8). Although the etiology of pressure sores is multifactorial (9), continuous pressure at the user seat interface is considered the most important factor (10,11). Therefore, wheelchair features are very important for posture and pressure sores. In our study, wheelchair features will be examined and these features will be compared with patient satisfaction. In addition, wheelchair characteristics and patient satisfaction in different patient groups (such as spinal cord injury, Multiple Sclerosis, Cerebrovascular Incident (stroke)) will also be discussed.

Hypotheses Ho: There is no difference between initial sitting pressure and posture in wheelchair users and sitting pressure and posture after 2 and 3 hours.

H1: There is a difference between the initial sitting pressure and posture in wheelchair users and the sitting pressure and posture after 2 and 3 hours.

H2: There is a difference between the initial sitting pressure and posture and the sitting pressure and posture after 2 and 3 hours in different patient groups.

H.4. Method: Individuals Patients who are being followed up in FTR or neurology Neurology clinics at Necmettin Erbakan University Meram Faculty of Medicine will be included in the study. In the G-Power analysis we conducted, Cascioli's study was based on comfort (12). However, we think that the number of people to be included in the study is low in terms of objectivity of the data. For this reason, a preliminary study will be conducted during the study and the sample number will be confirmed.

1. Physical characteristics and history taking: Patients will be asked in detail about age, height, weight, disease diagnosis and duration, and wheelchair characteristics.

   Inclusion criteria were:
   1. Patients with multiple sclerosis, myopathies, amyotrophic lateral sclerosis, polio and medulla spinalis incision,
   2. Being 18 years of age or older,
   3. have used a wheelchair for at least three months,
   4. being dependent on a wheelchair (all day) or at certain times of the day as the primary means of movement, Individuals will be excluded if they have suffered pressure sores within the last year.
2. Evaluations After taking the patient's history, the person was taken to MAT bed for 20 minutes. will be provided to rest. 20 minutes At the end, the patient who passes to the wheelchair will be asked to evaluate the comfort and discomfort they perceived after the first contact in the chair as 0 (none) -10 (very bad). Grading will be asked to evaluate the discomfort in the head, neck, back, waist, hips and legs, not the general sense of comfort. Meanwhile, pressure and posture will be evaluated.

   * Route-Reach test: This test is used to evaluate hamstring and trunk flexion flexibility. The subject will be asked to sit on the test table with both knees in extension on a firm surface and reach out with his hands and feet without bending the knees. The distance between the fingers and the tip of the test table is measured with a ruler

ELIGIBILITY:
Inclusion Criteria:

Patients with multiple sclerosis, myopathies, amyotrophic lateral sclerosis, polio and medulla spinalis incision, Being 18 years of age or older, have used a wheelchair for at least three months being dependent on a wheelchair as a primary mobility (all day) or at certain times of the day -

Exclusion Criteria:

Individuals will be excluded if they have suffered pressure sores within the past year.

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are being followed up in FTR or neurology Neurology clinics at Necmettin Erbakan University Meram Faculty of Medicine will be included in the study. In the G-Power analysis we conducted, the analysis was made based on comfort data in Cascioli's study (12). However, we think that the number of people to be included in the study is low in terms of objectivity of the data. For this reason, a preliminary study will be conducted during the study and the sample number will be determined.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Wheelchair First-Last Seating Pressure and Posture and Wheelchair Satisfaction | 45 minutes
  All af study
Sit-Reach test: Pressure Rating: It will be evaluated in kilograms | 2 two minutes
  the value will be recorded in centimeters (cm).
Pressure Rating | 3 minutes
  It will be evaluated in kilograms

SECONDARY OUTCOMES:
Evaluation of basic daily living activities (FIM) | 10 minutes
  The total FIM score can range from 18-126.
Craig Handicap Assessment and Reporting Technique (CHART) | 10 minutes
  Has a scale score ranging from 0 to 100
Wheelchair Skills Test (WST) for manual wheelchair users | 15 minutes
  Total WST Capacity Score = total of individual skill points / ([number of possible skills - number of NP points - number of TE points] x 3) X 100%
World Health Organization Quality of Life Scale (WHOQOL): | 5 minutes
  WHOQOL-BREF, unlike the long scale, consists of 4 domains. They do not have separate sections. This scale also has no total score. Each section and area scores a maximum of 20 points or 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Erdeo, Phd, Principal Investigator — Necmettin Erbakan Universİty; Sami Küçükşen, Prof., Study Director — Necmettin Erbakan Universİty

IPD SHARING:
Plan to Share IPD: Yes
When the research is published, I will share my data over Mendeley data sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year

REFERENCES:
- [Background] Ferrarin M, Andreoni G, Pedotti A. Comparative biomechanical evaluation of different wheelchair seat cushions. J Rehabil Res Dev. 2000 May-Jun;37(3):315-24. PMID 10917263
- [Result] Linder-Ganz E, Shabshin N, Itzchak Y, Gefen A. Assessment of mechanical conditions in sub-dermal tissues during sitting: a combined experimental-MRI and finite element approach. J Biomech. 2007;40(7):1443-54. doi: 10.1016/j.jbiomech.2006.06.020. Epub 2006 Aug 21. PMID 16920122
- [Result] Crenshaw RP, Vistnes LM. A decade of pressure sore research: 1977-1987. J Rehabil Res Dev. 1989 Winter;26(1):63-74. No abstract available. PMID 2645399
- [Result] Krause JS, Vines CL, Farley TL, Sniezek J, Coker J. An exploratory study of pressure ulcers after spinal cord injury: relationship to protective behaviors and risk factors. Arch Phys Med Rehabil. 2001 Jan;82(1):107-13. doi: 10.1053/apmr.2001.18050. PMID 11239295